CLINICAL TRIAL: NCT04290377
Title: A Study on the Effectiveness of Upper Extremity Rehabilitation Training Using Brain-Machine Interface Biofeedback in Stroke Patients With Hemiplegia
Brief Title: Upper Extremity Rehabilitation Training Using Brain-Machine Interface Biofeedback in Stroke Patients With Hemiplegia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to difficulties in recruiting the targeted number of participants and the departure of a key researcher responsible for bio-signal data processing.
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Nam-Jong Paik, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B-1908-559-301
Record Dates: First submitted 2020-02-25; First posted 2020-02-28 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Stroke; Hemiplegia
Keywords: Neural plasticity; Brain Machine Interface; Functional near-infrared spectroscopy; Stroke; Upper extremity; Function; Recovery
MeSH Terms: conditions — Stroke; Hemiplegia

STUDY DESIGN:
Intervention Model Description: Phase1 (chronic stroke): with-in group (one group) multiple measurements Phase2 (subacute stroke): Randomized controlled study. Control (OT plus OT) vs Experimental (OT plus BMI-assisted OT)
Who Masked: Investigator, Outcomes Assessor
Masking Description: Impossible to mask participants and care providers due to using a device that is so obvious.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional OT + Motor Imagery OT (Active Comparator): Conventional OT (30 minutes/day) plus Motor Imagery OT (30 minutes/day) for 10 days.
  Interventions: Other: Motor imagery OT
- Conventional OT + BMI-assisted Motor Imagery OT (Experimental): Conventional OT (30 minutes/day) plus BMI-assisted motor imagery OT (30 minutes/day) for 10 days.
  Interventions: Device: BMI-assisted motor imagery OT

INTERVENTIONS:
Device: BMI-assisted motor imagery OT — As the goal of the intervention is to promote finger extension in participants who are unable to extend his/her finger due to stroke, the pneumatic glove provides extension assist when appropriate brain activity is present. The brain activity is obtained by Functional Near-Infrared Spectroscopy (fNIRS). Hypothetically, this will repeatedly induce brain activation that is related to finger extension.
  Arms: Conventional OT + BMI-assisted Motor Imagery OT
Other: Motor imagery OT — In Motor imagery OT, Subjects try to extend their fingers (imagine) without BMI assistance. All other setting is equal to BMI-assisted motor imagery OT.
  Arms: Conventional OT + Motor Imagery OT

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of upper extremity rehabilitation using a Brain-Machine Interface (BMI) in individuals with hemiplegia due to stroke. The main questions it aims to answer are:

* Can BMI-assisted occupational therapy improve the Fugl Meyer Assessment-Upper Limb (FMA-UL) score in chronic stroke participants?
* How does the effectiveness of BMI-assisted occupational therapy compare to conventional occupational therapy alone?

Participants will:

Undergo 5 sessions of BMI-assisted occupational therapy in phase 1. Be randomly allocated to either a control group (receiving conventional occupational therapy) or an experimental group (receiving BMI-assisted OT plus conventional OT) in phase 2.

Researchers will compare the control group (OT plus OT) and the experimental group (BMI-assisted OT plus OT) to see if there is a significant difference in the change of FMA-UL score between the two groups.

DETAILED DESCRIPTION:
This is a study to evaluate the efficacy of upper extremity rehabilitation using Brain-Machine Interface (BMI) on individuals with hemiplegia due to stroke. BMI is a device that can record and analyze human brain signals (in this study Functional near-infrared spectroscopy was used) and also provide live feedback (by pneumatic glove movement) to the individual wearing it. This device hypothetically enables more accurate training by reinforcing the correctly activated brain signal repeatedly then conventional therapy.

In phase 1 study investigators will evaluate the feasibility of BMI on chronic stroke participants. 5 sessions of BMI-assisted occupational therapy (OT) will be performed and the Fugl Meyer Assessment-Upper Limb (FMA-UL) score change between the pre-treatment and post-treatment will be analyzed by paired t-test.

In phase 2 study, a randomized controlled study will be performed by randomly allocating participants to either control (OT plus OT) or experimental group (BMI-assisted OT plus OT) and the difference of FMA-UL score change between the two groups will be analyzed by Student's t-test.

ELIGIBILITY:
Inclusion Criteria:

* Subcortical stroke with hemiplegia
* 1st stroke
* Time since onset is less than 3 months
* Brunnstrom stage 2,3

Exclusion Criteria:

* Recurred stroke
* MMSE score below 10
* Delirium
* Unstable medical condition
* Pregnancy
* Cannot sustain sitting position for 30 minutes
* Pain that limits upper extremity exercise

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-13 (Actual)

PRIMARY OUTCOMES:
Change of Fugl Meyer Assessment-Upper Limb (FMA-UL) Score | Baseline evaluation (T0), Evaluation after 2 weeks of therapy (T1 [immediately or 1 day after treatment termination]), Evaluation after 1 month of T1 (T2), Evaluation after 3 month of T2 (T3).
  Impairment measurement

SECONDARY OUTCOMES:
Change of Finger Tapping Test Score (taps/minute) | Baseline evaluation (T0), Evaluation after 2 weeks of therapy (T1 [immediately or 1 day after treatment termination]), Evaluation after 1 month of T1 (T2), Evaluation after 3 months of T2 (T3).
  The number of finger tapping on I-pad screen per 10 seconds for 1 session. Total : 3 sessions
Change of Finger Extension (Metarcapophalangeal [MCP] joint) Range of Motion (degree) | Baseline evaluation (T0), Evaluation after 2 weeks of therapy (T1 [immediately or 1 day after treatment termination]), Evaluation after 1 month of T1 (T2), Evaluation after 3 month of T2 (T3).
  Range of motion of 2nd finger is measured with Goniometer.
Change of Hand grasp power (lb) | Baseline evaluation (T0), Evaluation after 2 weeks of therapy (T1 [immediately or 1 day after treatment termination]), Evaluation after 1 month of T1 (T2), Evaluation after 3 month of T2 (T3).
  Measured with Dynamometer
Change of Brunnstrom Stage | Baseline evaluation (T0), Evaluation after 2 weeks of therapy (T1 [immediately or 1 day after treatment termination]), Evaluation after 1 month of T1 (T2), Evaluation after 3 month of T2 (T3).
  Observational evaluation of the stage of recovery of a stroke patient. There are six stages (1: flaccid, 2: spasticity appears, 3: pronounced spasticity, 4: start of deviation from spasticity, 5: spasticity decreased more than 4 and complex movement combinations are possible, 6: No more spasticity present, near normal to normal movement
Change of muscle strength (Medical Research Council)-Upper extremity | Baseline evaluation (T0), Evaluation after 2 weeks of therapy (T1 [immediately or 1 day after treatment termination]), Evaluation after 1 month of T1 (T2), Evaluation after 3 month of T2 (T3).
  Manual measurement of muscle strength. Range from 0 to 5. When there is absolute no movement of muscle it scored as 0. When muscle activation is felt by palpation but no movement is present it is scored as 1. If full range of motion is possible with gravity removed it is scored as 2. If one can move his/her joint to full range of motion against gravity but without other resistance it is scored as 3. If one can resist mild resistance it is score as 4. If one's muscle strength is normal it is scored as 5.
Change of Box and Block Test (BBT) Score (boxes/60 second) | Baseline evaluation (T0), Evaluation after 2 weeks of therapy (T1 [immediately or 1 day after treatment termination]), Evaluation after 1 month of T1 (T2), Evaluation after 3 months of T2 (T3).
  An observational measurement on manual dexterity. The observer counts the number of boxes that participant can move across the mid-line dissection board in a limited time (60 seconds).
Change of Functional near-infrared spectroscopy Connectivity | Baseline evaluation (T0), Evaluation after 2 weeks of therapy (T1 [immediately or 1 day after treatment termination]), Evaluation after 1 month of T1 (T2), Evaluation after 3 months of T2 (T3).
  Near infrared spectroscopy is a tool that can measure the brain activity and subsequently analyze connectivity between each recording spot. The connectivity will be reported as an illustration or image
Change of Modified Ashworth Scale (MAS) of upper extremity | Baseline evaluation (T0), Evaluation after 2 weeks of therapy (T1 [immediately or 1 day after treatment termination]), Evaluation after 1 month of T1 (T2), Evaluation after 3 months of T2 (T3).
  Measures resistance during passive muscle stretching and is used as a simple measure of spasticity. 0: No increase in muscle tone, 1: Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension. 2: More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved. 3: Considerable increase in muscle tone, passive movement difficult. 4: Affected part(s) rigid in flexion or extension.
Change of range of motion of finger extension (degrees) measured with Camera and marker | Baseline evaluation (T0), Evaluation after 2 weeks of therapy (T1 [immediately or 1 day after treatment termination]), Evaluation after 1 month of T1 (T2), Evaluation after 3 months of T2 (T3).
  Markers (stickers) are placed on finger joints (Proximal phalangeal joint, Distal phalangeal joint) and finger tip of the 2nd finger. The camera will recognize the marker and measure the range of 2nd finger extension.

CONTACTS AND LOCATIONS:
Overall Officials: Nam-Jong Paik, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No